CLINICAL TRIAL: NCT00820287
Title: Identification of Predictive Markers for Testis Cancer in a Population of Men With High Risk
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APN 2004
Record Dates: First submitted 2009-01-09; First posted 2009-01-12 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2009-01

CONDITIONS: Testicular Cancer
Keywords: Testicular cancer; incidence; young men
MeSH Terms: conditions — Testicular Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Biopsy of testicular tumor — testicular biopsies performed through open surgery

SUMMARY:
Testis cancer with germ cells is the most frequent cancer of young men and its incidence is in constant increase in many industrialized countries, as in France. An increased risk of developing testis cancer has been described in patients with testicular ectopia history and testicular cancer history (controlateral testicular cancer) and more recently suggested in a population of hypofertile men with altered spermatogenesis. To a better understanding of this risk, an attempt of characterization of this group of patients has been proposed in the present work.

The general objective of this project is to characterize morphological and molecular markers of hypofertility which could serve as predictive markers of testis malignant transformation.

In this project conducted in 3 establishments, the investigators propose:

* To select a population of hypofertile patients exhibiting compatible clinical and morphological characters with a high risk of testis tumoral transformation (secretory azoospermia and/or a history of testicular ectopia. To determine the spermatogenic arrests on histological criteria (score of Jonhsen).
* To study the expression of four proteins or family of proteins suspected of being involved in testis tumorogenesis such as: the Placenta Alkaline Phosphatase (PLAPE), cyclin A1, VASA and connexin (Cx) by immunohistochemistry and by real-time quantitative RT-PCR analysis real-time analyses.
* To establish a possible correlation between the clinical data, spermatogenesis arrest and the expression of these biomarkers.

These approaches would allow to identify, in this population of hypofertile patients, subgroups of men who could develop tumours with germ cells, and subsequently to propose potential biomarkers for testis cancer. A more clinical observation of these subgroups will be also proposed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with infertility azoospermia
* Age 18 to 35 years
* Definition of clinical and biological character of azoospermia: testicular volume less than 10 ml and FSH more than 10 IU / l
* Normal karyotype
* Surgical exploration included in a standardized medical aid to procreation
* Testicular biopsy performed by traditional surgery
* Patient informed about the research protocol and having signed consent to conduct a further testicular biopsy included in this study.

Exclusion Criteria:

* adults protected by law, minors
* Individuals who are not affiliated to a social security
* Subjects hospitalized for any reason other than research.
* Patients will be used to support reproductive techniques:
* Positive serology (HIV, hepatitis ...).
* Patients with karyotype anomalies and unfavourable genetic counselling

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2005-09; Primary Completion 2009-01 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Analysis of 4 recognized tumorogenesis biomarkers in testicular biopsies of a population of hypofertiles men in theory supposed to present an increased incidence of testicular cancer development | 4 years

SECONDARY OUTCOMES:
Identification of spermatogenic achieving by conventional histology (analysis of Jonhsen's score) | 4 years
Establishment of one or more correlation (s) between the level of expression of biomarkers of tumorogenesis: Jonhsen score, the rate of circulating spermatogenesis serum markers (AMH, inhibin ...). | 4 years
Establishment of a correlation between the level of expression of of tumorogenesis testicular biomarkers, the presence of testicular microlithiasis and carcinoma in situ of the testis | 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France